CLINICAL TRIAL: NCT06170502
Title: Developing and Evaluating a Mobil Application for Rational Drug Use in Parents of Pediatric Patients After Discharge (Akilmobil)
Brief Title: Developing and Evaluating a Mobil Application AKILMOBIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayşegül Karaca, principal investigator, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TUBITAK 2023
Record Dates: First submitted 2023-09-01; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Survey Application
Keywords: drug; nurse; rational medicine

STUDY DESIGN:
Intervention Model Description: The type of study is a randomized controlled experimental study. In the research, it is aimed to evaluate the effectiveness of the mobile application (Akil Mobil).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mobile application development and implementation (Experimental): The aim of the project is to develop and evaluate the effectiveness of a mobile application (AkilMobil) that prevents parents who continue to use drugs for their children at home after their child is discharged from the hospital. The research is a randomized controlled experimental study. In the study, "The Form for Determining the Educational Needs of Parents Administering Medicines at Home", "Introductory Information Form", "Parental Drug Preparation Information Evaluation Form", "Parent Evaluation Form in Suspension Drug Administration", "Capsule Drug Application Parent Evaluation Form", developed by the researchers in line with the literature, "Tablet Pharmaceutical Application Parent Evaluation Form", "Mobile Application Usability Questionnaire", "AkilMobil Expert Opinion Evaluation Form" and "STAI State Anxiety Inventory" developed by Spielberger et al. will be used.
  Interventions: Device: Using the mobile application and applying the survey

INTERVENTIONS:
Device: Using the mobile application and applying the survey — In the study, "The Form for Determining the Educational Needs of Parents Administering Medicines at Home", "Introductory Information Form", "Parental Drug Preparation Information Evaluation Form", "Parent Evaluation Form in Suspension Drug Administration", "Capsule Drug Application Parent Evaluation Form", developed by the researchers in line with the literature, "Tablet Pharmaceutical Application Parent Evaluation Form", "Mobile Application Usability Questionnaire", "AkilMobil Expert Opinion Evaluation Form" and "STAI State Anxiety Inventory" developed by Spielberger et al. will be used.

SUMMARY:
The research was planned to develop the mobile application (Akil Mobil) that will be designed for parents who continue to use drugs for their children at home after their child is discharged from the hospital and after the discharge education is completed. The type of study is a randomized controlled experimental study.

DETAILED DESCRIPTION:
The irrational use of drugs is a major problem all over the world. About half of the patients cannot use the drugs correctly. Over, under or misuse of drugs leads to waste of resources and poor health conditions. The patients and their relatives who manage the use of drugs at home are most important componenets in this regard. Administration of the medication at home to the children mostly lead by parents.

Despite being informed during discharge, parents can make many mistakes in adjusting the dosage, preparing and administering tablet, capsule, suspension forms of drugs. And there are difficulties in accessing reliable sources of information.

It is necessary to keep the knowledge and skills of the parents of children with chronic diseases, who uses drugs for a long time, up-to-date. Therefore, continuous and accessible training and support systems are needed. Recently, mobile applications that can be easily accessed from mobile phones have become widespread thanks to technological developments. Regardless of their socioeconomic level, anyone with a smartphone can use these applications. A mobile application with home drug preparation and application can provide information and support for parents in the preparation and administration of appropriate doses.

For this reason, the aim of this project is to develop and evaluate a mobile application (AkilMobil) that prevents parents who continue to use drugs for their children at home after their child is discharged from the hospital. The research is a randomized controlled experimental study. In the study, "Education Needs of Parents who Administering Medicines at Home Form", "Descriptive Information Form", "Parental Drug Preparation Information Evaluation Form", " Suspension Drug Administration Parent Evaluation Form", "Capsule Drug Administration Parent Evaluation Form", "Tablet Drug Administration Parent Evaluation Form", "Mobile Application Usability Questionnaire", "AkilMobil Expert Opinion Evaluation Form" developed by the researchers in line with the literature, and "STAI State Anxiety Inventory" developed by Spielberger et al. will be used.

In the application, there will be drug information, indications, effects, side effects, preparation and administration methods, instructions for use, drug interaction information, dose calculation and drug preparation videos of drugs that are frequently used in chronic diseases, which are understood by parents. Interaction with users will be provided with frequently asked questions and the opportunity to ask researchers directly. With this application, parents can prevent dose errors due to lack of information while preparing drugs at home and information pollution due to applying to incorrect and insufficient sources. The mobile application's ease of access, presentation of visual resources and providing understandable information are the original values of our work. It is a technological advance for rational drug use and quality health care.

ELIGIBILITY:
Inclusion Criteria:

* Treating the disease condition and being discharged
* Continuing to use medication at home after discharge
* Parents should be able to speak and understand Turkish and be literate.
* Having an Android mobile phone for the mobile application
* Having the video call application on the mobile phone and accepting the video calling application to be made after 1 month
* Voluntary written and verbal informed consent has been obtained from the parents.

Exclusion Criteria:

* Parents' unwillingness to continue working at any stage of the research
* Termination of drug use due to the termination of their children's treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Mobile Application Usability Survey | 3 months
  Mothers with children with chronic diseases were evaluated with a mobile application usability survey, change in medication preparation activities in the 3rd month.

CONTACTS AND LOCATIONS:
Locations (1):
- Aysegul, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to the development